CLINICAL TRIAL: NCT01378767
Title: Biochemical, Hemodynamic, and Anthropometric Effects of a 21-day Daniel Fast in Men and Women
Brief Title: Health Benefits of a 21-day Daniel Fast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Dr. Richard Bloomer, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110184
Record Dates: First submitted 2011-06-10; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Effects of Krill Oil on Human Health
Keywords: Dietary restriction; oxidative stress; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Krill oil capsules (Active Comparator): Two grams per day daily for 21 days
  Interventions: Dietary Supplement: Krill oil supplementation
- Coconut oil capsules (Placebo Comparator): Two grams per day for 21 days
  Interventions: Dietary Supplement: Krill oil supplementation

INTERVENTIONS:
Dietary Supplement: Krill oil supplementation — During a 21-day Daniel Fast, group one supplemented with krill oil capsules (two grams per day) while group two supplemented with a placebo (coconut oil capsules at two grams per day).
  Other Names: Now Foods Neptune Krill Oil, 1000 mg- 60 Soft Gels; Brand NOW; Part Numbers 14431, 1627, 82048, NOW-01627, NWF-16270, NWF622; UPC 733739016270; Now Foods Coconut Oil, 1000 mg- 120 Soft Gels; Part Numbers 091363-2, 1718, 18918, 24230, 5933510, 6485, 71668, 806542, NWF-17185, NWF119; UPC 733739017185

SUMMARY:
The investigators hypothesized that individuals supplementing with krill oil capsules (two grams per day) would experience enhanced improvements in health-related variables during a 21-day Daniel Fast.

DETAILED DESCRIPTION:
One of the main purposes of the this investigation was to determine if krill oil supplementation (two grams per day for 21 days) enhances the effects of a 21-day Daniel Fast, particularly in regards to blood lipids and lipid peroxidation. The investigators were also interested in determining if adiponectin and/or resistin change in response to the fast, as these adipokines could potentially mediate the favorable glucoregulatory changes the investigators observed in our initial investigation of a 21-day Daniel Fast. Finally, the investigators sought to determine the changes in macronutrient and micronutrient intake during a Daniel Fast, and how these dietary changes affect our selected hemodynamic, anthropometric, blood lipid, glucoregulatory, oxidative stress, inflammatory, renal, and hepatic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must be willing to partake in a vegan diet for 21 days.
* Must be willing to consume either krill oil or coconut oil capsules (assigned randomly).

Exclusion Criteria:

* Smokers
* regular consumption of antioxidant supplements
* women who were pregnant or seeking to become pregnant
* poor veins (veins that made it difficult to successfully obtain a blood draw - this was determined via a visual inspection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood Lipids | Change from baseline at 3 weeks
  Total Cholesterol, LDL-C, HDL-C, VLDL-C, Triglyerides
Glucoregulatory markers | Change from baseline at 3 weeks
  Blood glucose, blood insulin, Serum resistin, serum adiponectin
Markers of Oxidative Stress and Antioxidant Status | Change from baseline at 3 weeks
  Plasma malondialdehyde, plasma hydrogen peroxide, plasma nitrate/nitrite, Trolox Equivalent Antioxidant Capacity (measured in serum)
Blood Pressure | Change from baseline at 3 weeks
  Systolic blood pressure, diastolic blood pressure
C-reactive protein | Change from baseline at 3 weeks

SECONDARY OUTCOMES:
Anthropometric Variables | Change from baseline at 3 weeks
  bodyweight, body mass index, waist circumference, hip circumference, body fat percentage, fat mass, fat free mass
Metabolic Panel | Change from baseline at 3 weeks
  Blood urea nitrogen, creatinine, sodium, potassium, carbon dioxide, calcium, protein, albumin, globulin, bilirubin, alkaline phosphatase, aspartate transaminase, alanine transaminase
Complete Blood Count | Change from baseline at 3 weeks
  White blood cells, red blood cells, hemoglobin, hematocrit, mean cell volume, mean cell hemoglobin, mean corpuscular hemoglobin concentration, red blood cell distribution width, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Bloomer, Doctorate, Principal Investigator — University of Memphis
Locations (1):
- Cardiorespiratory/Metabolic Laboratory, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Trepanowski JF, Kabir MM, Alleman RJ Jr, Bloomer RJ. A 21-day Daniel fast with or without krill oil supplementation improves anthropometric parameters and the cardiometabolic profile in men and women. Nutr Metab (Lond). 2012 Sep 13;9(1):82. doi: 10.1186/1743-7075-9-82. PMID 22971786